CLINICAL TRIAL: NCT01127360
Title: LUCAS. A Randomized, Prospective, Multicenter Study Comparing the Effect of Intravitreal Injection of Bevacizumab to Ranibizumab When Given to Patients With Neovascular Age-related Macular Degeneration
Brief Title: LUCAS (Lucentis Compared to Avastin Study)
Acronym: LUCAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1008
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: Anti-VEGF; Ranibizumab; Bevacizumab; exudative; macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Experimental): Bevacizumab 1,25 mg, intravitreal injections every 4th to 12th week
  Interventions: Drug: Bevacizumab; Drug: Ranibizumab
- Ranibizumab (Active Comparator): Ranibizumab 0,5 mg, intravitreal injection, every 4th to 12th week
  Interventions: Drug: Bevacizumab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Bevacizumab — Intravitreal injections
  Other Names: Avastin
Drug: Ranibizumab — Intravitreal injections
  Other Names: Lucentis

SUMMARY:
Age-related macular degeneration (AMD) is the most common cause of blindness in individuals over 50 years of age. Bevacizumab and ranibizumab are two agents developed by the American pharmaceutical corporation Genentech, both of which inhibit blood vessel growth factors. These drugs, when injected intraocularly, reduce the pathological growth of blood vessels in the macular area of the eye. Bevacizumab (Avastin) is an antibody developed for intravenous treatment of metastasized colon cancer. Ranibizumab (Lucentis) is an antibody fragment developed from a similar antibody. It was introduced 2006 as an effective treatment for wet AMD. Treatment costs are, however, up to 50 times higher compared to use of bevacizumab. Avastin has shown similar effects to ranibizumab, and has been used off-label in many countries, both before and after Lucentis received approval. There is thus a recognized need for large randomized studies to garner proper scientific proof of Avastin's effectiveness regarding exudative AMD.

LUCAS is a randomized multicenter study, performed in Norway, comparing ranibizumab and bevacizumab use for AMD. The goal of the study was to demonstrate if the two agents were equivalent regarding both efficacy and safety. A total of 441 patients with objective evidence of wet AMD were randomized to a double-blind treatment with ranibizumab or bevacizumab over the course of 2 years. The treatment interval was determined by a "Treat and Extend" protocol.

DETAILED DESCRIPTION:
LUCAS (LUcentis Compared to Avastin Study) A randomized, double-blind, prospective multicenter study comparing the effect of intravitreal injection of bevacizumab (Avastin) to ranibizumab (Lucentis) when given to patients with exudative (wet) age-related macular degeneration in Norway.

Version: 4, Protocol: 166-09, EudraCT: 2008-004225-41

Purpose:

LUCAS is a prospective, randomized, multicenter study comparing the effects of intravitreal injection of bevacizumab (Avastin) with ranibizumab (Lucentis) when given to patients with exudative (wet) AMD in Norway.

The study will include 420 patients to be recruited starting March 2009. The study will continue for 2 years after completed enrollment.

Design:

LUCAS is a multicenter, randomized, double-blind study, with 1:1 parallel groups treated with either bevacizumab (Avastin) 0.05 ml (25 mg/ml) or ranibizumab (Lucentis) 0,05 ml (10 mg/ml). The drug is injected intravitreally according to an "inject and extend" principle (5).

Randomization will be stratified by center and performed with minimization according to prognostic factors.

Treatment Regimen:

Bevacizumab (Avastin) will be given as an intravitreal injection of 0.05ml (25 mg/ml) from a vial containing 4 ml.

Ranibizumab (Lucentis) will be given as an intravitreal injection of 0.05 ml (10 mg/ml) from a vial containing 0.23 ml.

Follow-up and treatment will follow a principle called "inject and extend." This connotes the following: initial follow-up and injection with a 4 week intervals until the macula is dry. When dry, then follow-up and injection will be increased 2 weeks at a time. If the patient has a recurrence of wet AMD, then the interval is reduced by 2 weeks at a time until the macula is once again dry. The shortest interval is 4 weeks. When once again extending, the treatment interval shall not be as long as the interval of the original recurrence, as this could confer risk for new activity. Therefore further follow-up and injection occurs at the "ideal" interval which is hereby defined as being 2 weeks less than that of the original recurrence. With this method, the patient receives an injection at each follow-up, presuming that no complications occur. The maximum interval is limited to 12 weeks. Treatment will continue for 2 years. After the study is completed, then the patient is to be offered continued treatment, in accordance with the ophthalmology department's routines, If there is no response to treatment after 3 injections with a 4 week interval, then the patient shall be removed from the study and be offered alternative treatment, such as combination treatment with photodynamic therapy (PDT).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women.
2. Age ≥50 years.
3. Wet AMD in the study eye, defined as:

   Not previously treated active choroidal neovascular membrane (CNV), including retinal angiomatous proliferation (RAP), with edema involving the fovea as demonstrated with optical coherence tomography (OCT) and fluorescein angiography (FA). FA shall not be older than 7 days at randomization.

   Best corrected visual acuity (BCVA) in the study eye 20/25 - 20/320.
4. Only one eye of each study patient may be recruited into the study. If the non-study eye is being treated with intravitreal anti-VEGF therapy, or develops wet AMD, then the same drug being used in the study eye shall be used in the non-study eye. Treatment must be given double-blind in the non-study eye as well.

Exclusion Criteria:

1. Previous treatment of CNV in the study eye.
2. Participation in another AMD study, or use of other investigational medicines.
3. Anti-VEGF treatment in the non-study eye during the last 4 weeks.
4. Earlier or current treatment with systemic anti-VEGF drug.
5. Subretinal hemorrhage and/or fibrosis that involves ≥50 percent of the CNV lesion in the study eye.
6. CNV of other pathogenesis, such as pathologic myopia (defined as having a spherical equivalent of >8 diopters myopia) or Presumed Ocular Histoplasmosis Syndrome (POHS).
7. Presence of retinal diseases other than AMD (diabetic retinopathy, macular hole, etc) that lead to loss of visual acuity in the study eye.
8. Cataract that will presumably require operation within 2 years or other intraocular surgery or laser treatment during the last 3 months.
9. Impaired visualization of the retina (by vitreous hemorrhage, corneal dystrophy, etc.) that may hamper adequate diagnosis.
10. Intraocular pressure ≥25 mm Hg, measured before mydriasis, or uncontrolled glaucoma as evaluated by the examining ophthalmologist.
11. Active uveitis in the study eye or intraocular inflammation after use of Lucentis or Avastin in the non-study eye.
12. Infection in one or both eyes.
13. Premenopausal women who do not use appropriate birth control, or who are nursing.
14. Patients who for mental or physical reasons are unable to comply with the study's procedures,
15. Serious disease where there is a probability of death within the duration of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mean change in VA at 1 and 2 years as measured with the ETDRS chart | After 1 and 2 years
  Mean change in VA at 1 and 2 years as measured with the ETDRS chart (with a non-inferiority limit of 5 letters)

SECONDARY OUTCOMES:
Number of treatments. | After 1 and 2 years
  Number of treatments.
Proportion of patients losing fewer than 15 letters on ETDRS chart | After 1 and 2 years
  Proportion of patients losing fewer than 15 letters on ETDRS chart
Macular morphology as measured by FA and OCT after 2 years. | After 2 years
  Macular morphology as measured by FA and OCT after 2 years.
Adverse events | 2 years
  Frequency of ophthalmological and other health related adverse events during the 2 year study.
Number of non-responders. | After 2 years
  Number of non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Moan, Study Director — Director of Research at Oslo University Hospital; Ragnheidur Bragadottir, MD. PhD., Study Chair — Department of Ophthtalmology, Oslo University Hospital; Karina Berg, MD., Principal Investigator — Department of Ophthalmology, Oslo University Hospital; Terje Pedersen, Professor, Study Chair — Department of Preventative Medicine, Oslo University Hospital
Locations (1):
- Department of Ophthalmology, Oslo University Hospital, Oslo, Norway